CLINICAL TRIAL: NCT07187583
Title: Tapering of Biologics in Chronic Rhinosinusitis With Nasal Polyps
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Elizabeth M. Stevens, national coordinating investigator, and sub-investigator at Rigshospitalet, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-519758-35-01
Record Dates: First submitted 2025-09-11; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dosing of biological therapy (No Intervention): Continues dosing of mepolizumab (100 mg via injection pen, subcutaneous injection) or dupilumab (300 mg via injection pen, subcutaneous injection) every 4 weeks.
- Increased dosing interval of biological therapy (Active Comparator): Increases to a 6-week dosing interval at baseline - of mepolizumab (100 mg via injection pen, subcutaneous injection) or dupilumab (300 mg via injection pen, subcutaneous injection) - and if response to therapy is maintained, increases to 8-week dosing intervals at the follow-up visit in week 26. Thereafter, dosing every 8 weeks is maintained until the patient completes the trial at week 52.
  Interventions: Drug: increased dosing interval of biological therapy

INTERVENTIONS:
Drug: increased dosing interval of biological therapy — Increasing dosing interval of biological therapy for CRSwNP from every 4 weeks to every 6 weeks and if continued satisfactory response then to every 8 weeks.
  Arms: Increased dosing interval of biological therapy

SUMMARY:
The purpose of this study is to investigate the feasibility of extending the dosing intervals of biological therapies while maintaining optimal treatment effects in chronic rhinosinusitis with nasal polyps (CRSwNP).

DETAILED DESCRIPTION:
This is an investigator-initiated, independent, national multicenter study with a real-world design and Good Clinical Practice (GCP) monitoring. The study is a randomized controlled drug trial investigating the non-inferiority of extended dosing intervals compared with standard treatment for patients with CRSwNP receiving mepolizumab (100 mg) or dupilumab (300 mg) every 4 weeks. Approximately 135 patients will be enrolled from ear, nose and throat departments in all five regions of Denmark. The study duration is approximately 2.5 years, with each patient followed for 52 weeks.

Randomization At inclusion, patients are randomized 1:1 to the intervention or control group. Randomization is computer-based (REDCap).

Control group Continues dosing of mepolizumab or dupilumab every 4 weeks.

Intervention group Increases to a 6-week dosing interval at baseline, and if response to the biological therapy is maintained, increases to 8-week dosing intervals at the follow-up visit at week 26. Thereafter, dosing every 8 weeks is maintained until the patient completes the trial at week 52. In case of worsening of CRSwNP-related symptoms, the patient reverts to the last effective dosing interval.

Clinical visits Clinical follow-ups are conducted at weeks 0, 12, 26, 38, and 52. The visits at weeks 0, 26, and 52 are already planned as a standard part of biological treatment outside the protocol and include endoscopic rhinoscopy, smell testing, and questionnaires: Sinonasal Outcome Test 22 (SNOT-22), Work Productivity and Activity Impairment (WPAI), and Asthma Control Questionnaire (ACQ). The visits at weeks 12 and 38 are study-specific and include patient-reported symptom severity on a Visual Analogue Scale (VAS), endoscopic rhinoscopy, and completion of questionnaires (SNOT-22, WPAI).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Currently receiving treatment with either dupilumab (300 mg) or mepolizumab (100 mg) every four weeks.
* Having received the biologic at unchanged dosing interval for at least three months.
* For at least one year during treatment with biologics, the patients' CRSwNP must be categorized as "partly controlled" as defined by presence of 1-2 of the following seven items (also available in EPOS 2020 table in protocol):

  1. Nasal blockage: present on most days of the week
  2. Rhinorrhoea/postnasal drip: mucopurulent on most days of the week
  3. Facial pain/pressure: present on most days of the week
  4. Sense of smell: impaired
  5. Sleep disturbance or fatigue: present
  6. Nasal endoscopy: diseased mucosa
  7. Rescue treatment (systemic corticosteroids, ESS, antibiotics): need of 1 course of rescue treatment

of which 1-5 will be scored by the patient using VAS (0-10) and noted above 5.

Exclusion Criteria:

* Patients with excellent response to biologics (0 of the above-mentioned 7 items for partly controlled disease)
* Patients with no or limited response to biologics (>2 of the above-mentioned 7 items for partly controlled disease)
* Patients with a cancer diagnosis deemed by the investigator to preclude participation in the trial
* Patients who, because of language barriers, are not able to understand Danish written information and, thus, are not able to answer questionnaires
* Patients who currently receive biologics for any other disease (asthma not included)
* Patients who are not able to give informed consent (i.e., patients who are permanently incapable)
* Patients who are not eligible because of the investigator's judgement
* Patients who experience pregnancy during the study will be excluded after an unscheduled visit - active IVF treatment (please see below)
* Unwillingness to follow the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients achieving sustained partly controlled disease after tapering of biologics for CRSwNP | from enrollment (week 0) to week 52.
  "partly controlled" as defined by presence of 1-2 of the following 7 items:
  1. Nasal blockage: present on most days of the week
  2. Rhinorrhoea/postnasal drip: mucopurulent on most days of the week
  3. Facial pain/pressure: present on most days of the week
  4. Sense of smell: impaired
  5. Sleep disturbance or fatigue: present
  6. Nasal endoscopy: diseased mucosa
  7. Rescue treatment (systemic corticosteroids, ESS, antibiotics): need of 1 course of rescue treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Buchwald, MD, DMSc, prof., Study Director — Rigshospitalet, Dept. of Otorhinolaryngology, Head and Neck Surgery & Audiology
Locations (9):
- Denmark (9):
  - Dept of otorhinolaryngology, Aalborg University Hospital, Aalborg
  - Dept of otorhinolaryngology, head and neck surgery, Aarhus University Hospital, Aarhus
  - Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Copenhagen University, Rigshospitalet, Copenhagen
  - Esbjerg Og Grindsted Sygehus, Esbjerg
  - Dept of otorhinolaryngology, Gødstrup Regional Hospital, Herning
  - Dept of otorhinolaryngology, Nordsjaellands Hospital, Hillerød
  - Dept of otorhinolaryngology, Sjællands Universitetshospital, Køge
  - Dept of otorhinolaryngology, Odense University Hospital, Odense
  - Dept of otorhinolaryngology, Lillebaelt Hospital, Vejle

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT07187583/Prot_SAP_000.pdf